CLINICAL TRIAL: NCT00590187
Title: A Randomized Phase 2 Study of Oral Sapacitabine in Elderly Patients With Acute Myeloid Leukemia Previously Untreated or in First Relapse, or Previously Treated Myelodysplastic Syndromes
Brief Title: Efficacy Study of Oral Sapacitabine to Treat Acute Myeloid Leukemia in Elderly Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYC682-06
Record Dates: First submitted 2007-12-23; First posted 2008-01-10 (Estimated); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — sapacitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- A sapacitabine (Experimental): 200 mg b.i.d. x 7 days every 3-4 weeks
  Interventions: Drug: Sapacitabine, Arm A
- B sapacitabine (Experimental): 300 mg b.i.d. x 7 days every 3 - 4 weeks
  Interventions: Drug: Sapacitabine, Arm B
- C sapacitabine (Experimental): 400 mg b.i.d. x 3 days/week x 2 weeks every 3 - 4 weeks
  Interventions: Drug: Sapacitabine, Arm C
- D sapacitabine (Experimental): 200 mg b.i.d. x 7 consecutive days every 4 weeks
  Interventions: Drug: Sapacitabine, Arm D
- E sapacitabine (Experimental): 300 mg q.d. x 7 consecutive days every 4 weeks
  Interventions: Drug: sapacitabine, Arm E
- F sapacitabine (Experimental): 300 mg b.i.d. x 3 consecutive days per week for 2 weeks every 4 weeks
  Interventions: Drug: sapacitabine, Arm F
- G sapacitabine (Experimental): 200 mg b.i.d. x 7 consecutive days every 4 weeks
  Interventions: Drug: Sapacitabine, Arm G
- H sapacitabine (Experimental): 300 mg q.d. x 7 consecutive days every 4 weeks
  Interventions: Drug: Sapacitabine, Arm H
- I sapacitabine (Experimental): 100 mg q.d. x 5 consecutive days per week for 2 weeks every 4 weeks
  Interventions: Drug: Sapacitabine, Arm I

INTERVENTIONS:
Drug: Sapacitabine, Arm A — 200 mg b.i.d. x 7 days every 3-4 weeks
  Other Names: CYC682
  Arms: A sapacitabine
Drug: Sapacitabine, Arm B — 300 mg b.i.d. x 7 days every 3 - 4 weeks
  Other Names: CYC682
  Arms: B sapacitabine
Drug: Sapacitabine, Arm C — 400 mg b.i.d. x 3 days/week x 2 weeks every 3 - 4 weeks
  Other Names: CYC682
  Arms: C sapacitabine
Drug: Sapacitabine, Arm D — 200 mg b.i.d. x 7 consecutive days every 4 weeks
  Other Names: CYC682
  Arms: D sapacitabine
Drug: sapacitabine, Arm E — 300 mg q.d. x 7 consecutive days every 4 weeks
  Other Names: CYC682
  Arms: E sapacitabine
Drug: sapacitabine, Arm F — 300 mg b.i.d. x 3 consecutive days per week for 2 weeks every 4 weeks
  Other Names: CYC682
  Arms: F sapacitabine
Drug: Sapacitabine, Arm G — 200 mg b.i.d. x 7 consecutive days every 4 weeks
  Other Names: CYC682
  Arms: G sapacitabine
Drug: Sapacitabine, Arm H — 300 mg q.d. x 7 consecutive days every 4 weeks
  Other Names: CYC682
  Arms: H sapacitabine
Drug: Sapacitabine, Arm I — 100 mg q.d. x 5 consecutive days per week for 2 weeks every 4 weeks
  Other Names: CYC682
  Arms: I sapacitabine

SUMMARY:
The objective is to treat elderly AML and MDS patients with sapacitabine.

DETAILED DESCRIPTION:
The main objective of this study is to learn which sapacitabine treatment is more likely to keep the cancer in check for at least one year in AML patients who are at least 70 years of age or older and in MDS patients who are at least 60 years of age.

ELIGIBILITY:
Inclusion Criteria:

* A histologically or pathologically confirmed diagnosis of AML based on WHO classification which is previously untreated by systemic therapy or is in first relapse after achieving a complete remission to initial induction, consolidation and/or maintenance therapy or MDS with IPSS scores of intermediate -2 or higher risk risk which has been previously treated with hypomethylating agents
* Age 70 years or older for AML and 60 years or older for MDS
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate renal function defined as serum creatinine equal to or less than 1.5 x upper limit of normal (ULN)
* Adequate liver function defined as total bilirubin or direct bilirubin equal to or less than 1.5 x ULN; alanine aminotransferase (ALT or SGPT) equal to or less than 2.5 x ULN (5 x ULN if tumor has affected the liver)
* Life expectancy reasonably adequate for evaluating the treatment effect
* Patient must be able to swallow capsules
* Patients must be at least 2 weeks from prior systemic therapy, radiation therapy, major surgery, or other investigational therapy, and have recovered from clinically significant toxicities of these prior treatments
* All men and women of reproductive potential must agree to practice effective contraception for 4 weeks prior to study entry, during the entire study period and for one month after the study unless documentation of infertility exists
* Ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* AML is of the sub-type of acute promyelocytic leukemia
* Having received more than one induction systemic therapy for AML or having received a standard dose or high dose ara-C containing regimen for MDS
* Patients with known central nervous system (CNS) involvement by leukemia
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, active cancer(s) other than AML, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patients receiving intravenous antibiotics for infections that are under control may be included in this study
* Known to be HIV-positive

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M Kantarjian, MD, Study Chair — M.D. Anderson Cancer Center
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Division of Hematology-Oncology, Los Angeles, California
  - Stanford Hospitals and Clinics, Stanford, California
  - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institiute, Buffalo, New York
  - New York Medical College, Hawthorne, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt U Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kantarjian H, Faderl S, Garcia-Manero G, Luger S, Venugopal P, Maness L, Wetzler M, Coutre S, Stock W, Claxton D, Goldberg SL, Arellano M, Strickland SA, Seiter K, Schiller G, Jabbour E, Chiao J, Plunkett W. Oral sapacitabine for the treatment of acute myeloid leukaemia in elderly patients: a randomised phase 2 study. Lancet Oncol. 2012 Nov;13(11):1096-104. doi: 10.1016/S1470-2045(12)70436-9. Epub 2012 Oct 15. PMID 23075701
- See also: Oral sapacitabine for the treatment of acute myeloid leukaemia in elderly patients: a randomised phase 2 study. — https://doi.org/10.1016/S1470-2045(12)70436-9

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arms D through I were terminated prematurely because of financial restrictions. Accordingly the company made the determination of the dosing schedule which was used in the subsequent Phase 3 study based on the results of Arms A through C.
Period: Overall Study
Arm/Group | A Sapacitabine | B Sapacitabine | C Sapacitabine
Started | 40 | 20 | 45
Completed | 40 | 20 | 45
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Sapacitabine | B Sapacitabine | C Sapacitabine | Total
Number analyzed (Participants) | 40 | 20 | 45 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 40 | 20 | 45 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 7 | 20 | 44
  Male | 23 | 13 | 25 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 37 | 19 | 38 | 94
  Black | 1 | 1 | 3 | 5
  Hispanic | 2 | 0 | 4 | 6
Patients aged 70 years or higher [Count of Participants; unit: Participants] | 40 | 20 | 45 | 105

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Percentage of patients alive for one year measured from the date of randomization
Time Frame: up to 12 months from date of randomization
Population: Arms D through I were terminated prematurely because of financial restrictions. Accordingly the company made the determination of the dosing schedule which was used in the subsequent Phase 3 study based on the results of Arms A through C.
Measure: Number (95% Confidence Interval); unit: percentage of patients alive for one yea
Arm/Group | A Sapacitabine | B Sapacitabine | C Sapacitabine
Number analyzed (Participants) | 20 | 20 | 20
percentage of patients alive for one yea | 35 [16 to 59] | 10 [2 to 33] | 30 [13 to 54]

2. Secondary Outcome: CR and CRp
Description: Complete remission and complete remission without blood count recovery, transfusion requirements, hospitalized days and safety
Time Frame: From date of randomization until study withdrawal or death assessed up to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A Sapacitabine | B Sapacitabine | C Sapacitabine
Number analyzed (Participants) | 40 | 20 | 45
Participants | 6 | 2 | 8

ADVERSE EVENTS:
Time Frame: Median length of follow-up was 143 weeks.
Description: The definitions of adverse event and serious adverse event are in congruence with clinicaltrials.gov standard definitions. Arms D through I were terminated prematurely because of financial restrictions. Accordingly the company made the determination of the dosing schedule which was used in the subsequent Phase 3 study based on the results of Arms A through C.
Arm/Group | A Sapacitabine | B Sapacitabine | C Sapacitabine
All-Cause Mortality (participants affected / at risk) | 8/40 | 6/20 | 4/45
Serious Adverse Events (participants affected / at risk) | 40/40 | 20/20 | 45/45
Other Adverse Events (participants affected / at risk) | 40/40 | 20/20 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Sapacitabine (N=40) | B Sapacitabine (N=20) | C Sapacitabine (N=45)
Anemia (Blood and lymphatic system disorders) | 8 (8) | 12 (12) | 15 (15)
Febrile Neutropenia (Blood and lymphatic system disorders) | 16 (16) | 9 (9) | 22 (22)
Neutropenia (Blood and lymphatic system disorders) | 14 (14) | 10 (10) | 11 (11)
Throbocytopenia (Blood and lymphatic system disorders) | 24 (24) | 12 (12) | 22 (22)
Atrial fibrilation (Cardiac disorders) | 2 (2) | 2 (2) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1) | 4 (4)
Peripheral Oedema (General disorders) | 1 (1) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 5 (5) | 2 (2) | 5 (5)
Cellulitis (General disorders) | 3 (3) | 3 (3) | 5 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (6) | 13 (13)
Sepsis (General disorders) | 9 (9) | 3 (3) | 2 (2)
Anorexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3)
Arthralgia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (General disorders) | 0 (0) | 0 (0) | 3 (3)
Insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (General disorders) | 2 (2) | 0 (0) | 2 (2)
Epistaxis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (General disorders) | 1 (1) | 1 (1) | 1 (1)
Petechiae (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Hypotension (General disorders) | 2 (2) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Sapacitabine (N=40) | B Sapacitabine (N=20) | C Sapacitabine (N=45)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 4 (4)
Atrial fibrilation (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Abdominal pain (General disorders) | 6 (6) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (10) | 8 (8) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 23 (23) | 11 (11) | 17 (17)
Nausea (General disorders) | 16 (16) | 6 (6) | 23 (23)
Stomatitis (General disorders) | 4 (4) | 2 (2) | 7 (7)
Vomiting (General disorders) | 12 (12) | 5 (5) | 11 (11)
Fatigue (General disorders) | 19 (19) | 10 (10) | 13 (13)
Peripheral Oedema (General disorders) | 5 (5) | 8 (8) | 15 (15)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Fever (General disorders) | 6 (6) | 1 (1) | 9 (9)
Bacteraemia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Cellulitis (General disorders) | 3 (3) | 0 (0) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Anorexia (General disorders) | 9 (9) | 5 (5) | 8 (8)
Weight decrease (General disorders) | 3 (3) | 4 (4) | 3 (3)
Hypokalemia (Renal and urinary disorders) | 3 (3) | 0 (0) | 4 (4)
Arthralgia (General disorders) | 7 (7) | 0 (0) | 5 (5)
Back Pain (General disorders) | 4 (4) | 1 (1) | 6 (6)
Musculoskeletal chest pain (General disorders) | 1 (1) | 0 (0) | 6 (6)
Pain in extremity (General disorders) | 7 (7) | 1 (1) | 8 (8)
Dizziness (General disorders) | 7 (7) | 3 (3) | 10 (10)
Headache (General disorders) | 7 (7) | 0 (0) | 6 (6)
Insomnia (General disorders) | 4 (4) | 1 (1) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3) | 6 (6)
Dyspnoea (General disorders) | 15 (15) | 2 (2) | 10 (10)
Epistaxis (General disorders) | 6 (6) | 3 (3) | 5 (5)
Ecchymosis (General disorders) | 4 (4) | 3 (3) | 1 (1)
Petechiae (General disorders) | 4 (4) | 3 (3) | 7 (7)
Alopecia (General disorders) | 7 (7) | 2 (2) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 7 (7)
Hypotension (General disorders) | 4 (4) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-06-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT00590187/Prot_SAP_000.pdf